CLINICAL TRIAL: NCT01459887
Title: An Open-labeled, Multi-center, Randomized, Prospective Phase III Study Comparing CMAB304 in Combination With CHOP to CHOP Alone With CMAB304 Maintenance in Patients With DLBCL
Brief Title: Study of Recombinant Human-Mouse Chimeric Anti-CD20 Monoclonal Antibody to Treat Non-hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai CP Guojian Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 304NHL-050617
Record Dates: First submitted 2011-10-18; First posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: untreated, CD20-positive
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination group (Experimental)
  Interventions: Drug: CHOP combined with CMAB304
- sequential group (Experimental)
  Interventions: Drug: CHOP, CMAB304

INTERVENTIONS:
Drug: CHOP combined with CMAB304 — Patients treated with CHOP-304 undergo 1 cycle every 3 weeks, received CMAB304 at a dose of 375 mg/m2 on day 1 and CHOP on day 2 of each of the 6 cycles.
  Other Names: cyclophosphamide, doxorubicin, vincristine, prednisone
  Arms: combination group
Drug: CHOP, CMAB304 — First standard CHOP, then sequential CMAB304 in patients who reached a complete response or undocumented complete response at the end of treatment of 6 cycles.
  Other Names: cyclophosphamide, doxorubicin, vincristine, prednisone
  Arms: sequential group

SUMMARY:
CD20, the protein which is expressed on the surface of all mature B cells, is active in many B-cell lymphomas that express this molecule such as Diffuse Large B Cell Lymphoma (DLBCL), the most frequently occurring subtype of non-Hodgkin lymphomas. In clinical practice, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone combination chemotherapy (CHOP) is still considered one of the standard treatment to DLBCL. CMAB304(Retuxira), the chimeric monoclonal antibody is designed to targeted against CD20 for treatment of lymphoma diseases. This trial aimed to observe the safety and efficacy of CMAB304, by added CMAB304 to CHOP chemotherapy regimen compared with CHOP chemotherapy alone.

DETAILED DESCRIPTION:
Rituximab, a chimeric anti-CD20 monoclonal antibody, has been proved valuable treatment for CD20-positive DLBCL. The combination of rituximab with CHOP has been shown to increase both survival and response rate, in comparison to CHOP alone. CMAB304(Retuxira), a biosimilar of rituximab, was developed by Shanghai CP Guojian Pharmaceutical Co.,Ltd. Previous Phase I study showed that CMAB304 was well tolerated as monotherapy and the pharmacokinetic data exhibited a non-linear profile over the dose range of 250 to 500 mg/m2. In this study, efficacy and safety of CMAB304 were evaluated in DLBCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 70 year, male or female
2. Previously untreated
3. DLBCL patients with CD20-positive
4. Lymphoma lesions can be Measured and evaluated; Spiral CT or MR evaluation of the lesion must be ≥ 1cm; Measured by clinical examination or others must be ≥ 2cm
5. Normal blood test, adequate liver and renal function;
6. ECOG score 0~2
7. Life expectancy of greater than 3 months
8. No other malignancy treatment history, except cured carcinoma in situ of the cervix or squamous cell or basal cell skin cancer
9. Signed ICF

Exclusion Criteria:

1. DLBCL transformed from other low-grade NHL types
2. Primary central nervous system lymphoma, or primary gastrointestinal DLBCL
3. History of foreign protein allergies
4. Abnormal liver and/or renal function
5. Suspected or diagnosed central nervous system violation
6. Serious infection or organic diseases
7. Heart disease, heart failure, heart block above second degree, myocardial infarction occurred within six months
8. Breastfeeding or pregnant
9. Leukemia crisis or bone marrow metastases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
overall response rate | up to 18 weeks
  Tumor responses were assessed after 6 cycles of CMAB304-CHOP or 6 cycles of CHOP alone and classified as CR,CRu,PR,SD or PD.

SECONDARY OUTCOMES:
event-free survival | From date of randomization until the date of first documented progression or relapse, institution of a new anticancer treatment, or death from any cause, whichever came first, assessed up to 50 months
  Events were defined as disease progression or relapse, institution of a new anticancer treatment, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, PhD, Principal Investigator — Peking University Cancer Hospital & Institute; Daobin Zhou, PhD, Principal Investigator — Peking Union Medical College Hospital; Weijing Zhang, PhD, Principal Investigator — Affiliated Hospital of Chinese PLA Military Academy of Medical Sciences; Yiping Zhang, PhD, Principal Investigator — Zhejiang Cancer Hospital; Jifeng Feng, PhD, Principal Investigator — Jiangsu Cancer Institute & Hospital; Yu Yang, PhD, Principal Investigator — Fujian Cancer Hospital; Qitao Yu, PhD, Principal Investigator — Cancer Hospital of Guangxi Medical University; Yuankai Shi, PhD, Principal Investigator — Cancer Institute ＆Hospital. China Academy of Medical Sciences; Lugui Qiu, PhD, Principal Investigator — Tianjin Hematonosis Hospital; Ting Liu, PhD, Principal Investigator — West China Hospital; Wenbin Qian, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University; Ping Zou, PhD, Principal Investigator — Union Hospital of Tongji Medical College of Huazhong University of Science ＆ Technology; Zhongzhen Guan, PhD, Study Chair — Sun Yat-sen University; Huiqiang Huang, PhD, Study Director — Sun Yat-sen University
Locations (1):
- SUN-YAT-SEN university cancer center, Guangzhou, Guangdong, China